CLINICAL TRIAL: NCT06836973
Title: Efficacy and Safety of Blinatumomab for Treatment of Refractory Myasthenia Gravis.
Brief Title: Blinatumomab for Treatment of Refractory Myasthenia Gravis
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Da, Yuwei, M.D. (Individual)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LYS[2024]408-002
Record Dates: First submitted 2025-02-16; First posted 2025-02-20 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2025-02

CONDITIONS: Myasthenia Gravis
MeSH Terms: conditions — Myasthenia Gravis | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Blinatumomab (Experimental)
  Interventions: Drug: Blinatumomab

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is used at its starting dose of 9 µg per day and administered as continuous infusion for 5 days (total dose of 38.5 µg). After a 1-week pause, the patients receive a second 5-day infusion with blinatumomab of total 38.5 µg of the drug.

SUMMARY:
The goal of this clinical trial is to evaluate the efficacy and safety of Blinatumomab in the treatment of refractory myasthenia gravis, with the expectation of offering a new therapeutic option for refractory patients. The main questions it aims to answer are:

* Does Blinatumomab improve patients' clinical symptoms?
* Is Blinatumomab safe for the treatment of myasthenia gravis?

Participants will:

* Receive two cycles of intravenous Blinatumomab infusion, each lasting 5 days, with a 1-week interval between cycles.
* Visit the clinic once every 4 weeks for checkups and tests.
* Keep a diary of their symptoms and the types and dosages of medications.

ELIGIBILITY:
Inclusion Criteria:

* Age at onset > 18 years old
* The diagnosis of MG was based on the presence of typical myasthenic symptoms and supported by positive autoantibodies, electrophysiological studies, and/or the neostigmine test.
* Positive or negative for anti-AChR, and/or anti-MuSK, and/or anti-LRP4 antibodies.
* Refractory myasthenia gravis (MG) patients are defined as those who meet any of the following criteria: For patients with ocular MG, the condition is defined as having no significant improvement in disease symptoms (QMG score improvement <25%) after adequate dosing and duration of existing immunosuppressive drugs and targeted biologics, with no change or worsening in the post-intervention status (PIS), or if the PIS improves but disease symptoms worsen or relapse during the regular tapering of immunosuppressive treatment, severely affecting daily quality of life. For generalized MG, the patient must meet the following conditions: no improvement or worsening in PIS after adequate dosing and duration of existing immunosuppressive drugs and targeted biologics; improvement in PIS, but with an MG-ADL score ≥6 persisting for at least six months; remission or improvement in PIS, but with ≥2 episodes of disease exacerbation (MG-ADL ≥6) per year during tapering of immunotherapy medications; patients who, after experiencing a myasthenic crisis, undergo multiple immunotherapies including intravenous efgartigimod, eculizumab, immunoglobulin, plasma exchange, and high-dose intravenous methylprednisolone, and active infection control, but still cannot be weaned off the ventilator due to respiratory muscle weakness from MG for more than 14 days. (Note: This includes patients who cannot tolerate existing treatment drugs due to contraindications, comorbidities, or adverse drug reactions.)
* Receiving stable doses of medication prior to enrollment
* Written informed consent

Exclusion Criteria:

* Patients who have thymoma or have undergone thymectomy within six months
* Patients who have used other biologics prior to enrollment that may affect the efficacy assessment of blinatumomab.
* Severe cardiovascular, hepatic, renal, respiratory, or endocrine diseases, malignancies, or uncontrolled acute or chronic infections
* Pregnancy or lactation, unwillingness to avoid pregnancy
* Patients with other diseases that may affect the assessment of muscle strength
* Other conditions that would preclude participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2025-04-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Change of Myasthenia Gravis Activities of Daily Living (MG-ADL) Score from baseline | From baseline to 6 months
  The MG-ADL scale is an 8-item questionnaire. It is completed by trained interviewers based on the patients' subjective responses. The total score ranges from 0 to 24, with higher scores indicating greater impact of the disease on daily living activities.

SECONDARY OUTCOMES:
Change of Quantitative Myasthenia Gravis (QMG) Scores from baseline | From baseline to 6 months
  The QMG scale is a 13-item scale used to objectively assess muscle strength and fatigue in patients with myasthenia gravis. The total score ranges from 0 to 39, with higher scores indicating greater disease severity.
Time to achievement of minimal symptom expression (MSE) | From baseline to 6 months
  The MSE is a quantifiable, patient-reported outcome measure that assesses treatment goals in myasthenia gravis. It is defined as achieving an MG-ADL score of ≤1, indicating that clinical symptoms of MG are at their minimal level.
Change of Myasthenia Gravis Quantity-of-Life Scale (MG-QoL15) from baseline | From baseline to 6 months
  The MG-QOL15 scale is a 15-item questionnaire designed to assess the impact of myasthenia gravis on patients' daily life, physical function, social well-being, and mental health. The total score ranges from 0 to 60, with higher scores indicating poorer quality of life.
Change of Myasthenia Gravis Composite (MGC) scores from baseline | From baseline to 6 months
  The MGC scale is a 10-item scale that combines patient self-assessment and physician examination results. Each item is assigned a weight based on factors such as health risks, quality of life, and prognosis. The total score of the scale is 50 points, with higher scores indicating more severe disease.
Change of antibody titers from baseline | From baseline to 6 months
  MG antibodies are detected at enrollment and the titers of antibodies will be monitored monthly.
Treatment-Related Adverse Events (AEs) | From baseline to 6 months
  Record all AEs reported by patients during the study period.